CLINICAL TRIAL: NCT03253458
Title: In-vivo Focal Prostate Imaging With Confocal Laser Endomicroscopy and Optical Coherence Tomography
Brief Title: Focal Prostate Imaging With CLE and OCT
Acronym: FPI
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Collaborators: Amsterdam UMC, location VUmc (Other)
Responsible Party: Principal Investigator, Dr. T.M. de Reijke, Theo M. de Reijke, Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: NL57326.018.17; METC 2017_130 (Other: AMC-UvA)
Record Dates: First submitted 2017-08-07; First posted 2017-08-18 (Actual); Last update posted 2019-01-18 (Actual); Status verified 2019-01

CONDITIONS: Prostate Cancer
Keywords: Optical coherence tomography; Confocal Laser Endomicroscopy; Histology
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Tomography, Optical Coherence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Optical imaging (Experimental): All consenting patients will undergo Confocal Laser Endomicroscopy or Optical Coherence Tomography imaging prior to biopsy or surgery.
  Interventions: Device: Confocal Laser Endomicroscopy

INTERVENTIONS:
Device: Confocal Laser Endomicroscopy — Transperineal confocal laser endomicroscopy or optical coherence tomography measurements. Probe will be placed guided by ultrasound, similar procedure as transperineal template guided mapping biopsies.
  Other Names: Optical Coherence Tomography

SUMMARY:
The current limitations in prostate cancer diagnostics lead to over- and undertreatment for a significant fraction of patients. Confocal Laser Endomicroscopy (CLE) and Optical Coherence Tomography (OCT) are focal imaging modalities with potential for in-vivo prostate imaging. The investigators anticipate that integrating focal imaging with MRI/TRUS fusion will further improve prostate cancer detection and provides a real-time histopathological threedimensional representation of the tumor lesions.

This is an investigator-initiated, prospective in-vivo safety and feasibility study with transperineal template mapping biopsies (TTMB) and two focal imaging methods, CLE and OCT, in prostate tissue.

DETAILED DESCRIPTION:
Study design:

This is an investigator-initiated, prospective in-vivo safety and feasibility study with two procedures.

Procedure 1 (AMC):

Patients that are indicated for transperineal template mapping biopsies (TTMB) are included for procedure 1 and will receive transperineal CLE or OCT measurements prior to TTMB. Procedure 1 is to test the technical feasibility and safety of in-vivo focal imaging with CLE and OCT. Only if transperineal CLE or OCT measurements are possible, the investigators proceed with procedure 2.

For procedure 1: 4 patients that are scheduled for TTMB; 2 patients for CLE and 2 patients for OCT.

Procedure 2 (VUmc):

Patients scheduled for a robot-assisted laparoscopic prostatectomy (RALP) will be included in procedure 2 and receive transperineal CLE or OCT measurements prior to their surgery. Results will be correlated with histology by correlating biopsies during the TTMB procedure or with RALP the measurement trajectory will be marked. After the RALP, the prostate will be cut exactly through the measurement trajectory for whole mount coupes. In high-risk of high-intermediate-risk patients receiving an extended pelvic lymph node dissection with the RALP, ex-vivo CLE measurements will be performed.

For procedure 2: 10 patients that are scheduled for RALP; 5 patients for CLE and 5 patients for OCT. Intervention: Transperineal CLE or OCT measurements will be performed directly prior to the TTMB or RALP. The CLE and OCT probes are inserted by a needle with the same diameter as a biopsy gun. In the case of RALP, measurement trajectories will be marked for histopathology correlation.

Intervention:

Transperineal CLE or OCT measurements will be performed directly prior to the TTMB or RALP. The CLE and OCT probes are inserted by a needle with the same diameter as a biopsy gun. In the case of RALP, measurement trajectories will be marked for histopathology correlation.

ELIGIBILITY:
Inclusion criteria

* age ≥ 18 years
* signed informed consent
* mpMRI data available

Exclusion criteria

* Patients with a known allergic reaction to fluorescein cannot participate in this study.
* Documented acute prostatitis or urinary tract infections
* No ability to stop anticoagulant or antiplatelet therapy
* Medical history of a bleeding disorder or if available platelet Count <140/uL, prothrombin time >14.5 sec., partial thromboplastin time >34 sec.
* Major concurrent debilitating illness or ASA ≥4
* Biological or chemotherapy for PCa
* Hormonal therapy within last six months
* Has any medical condition or other circumstances which would significantly decrease the chances of obtaining reliable data, achieving study objectives, or completing the study
* Is incapable of understanding the language in which the information for the patient is given

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Prostate cancer only occurs in male
Enrollment: 14 (Estimated)
Dates: Start 2018-05-11 (Actual); Primary Completion 2019-12-31 (Estimated); Study Completion 2020-07-01 (Estimated)

PRIMARY OUTCOMES:
Visual image criteria for CLE and quantitative parameters (attenuation coefficient and residue) of OCT for the characterization of the prostate tissue | 2 years
  * Describing visual characteristics on CLE imaging
  * Attenuation coefficient on OCT imaging calculated with our in-house build software
  * Residue of the OCT imaging calculated with our in-house build software

SECONDARY OUTCOMES:
Technical feasibility of CLE and OCT imaging in the prostate by a transperineal approach | 2 years
  * Tissue visualization is not blocked by blood on CLE and OCT imaging
  * OCT image quality determination by visibility in depth
Safety of CLE and OCT imaging in the prostate | 2 years
  Procedure-related adverse events of needle based CLE and OCT

CONTACTS AND LOCATIONS:
Overall Officials: Theo M de Reijke, MD, Principal Investigator — AMC-UvA
Locations (1):
- AMC University Hospital, Amsterdam, North Holland, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] van Riel LAMJG, Swaan A, Mannaerts CK, van Kollenburg RAA, Savci Heijink CD, de Reijke TM, de Bruin DM, Freund JE. Image-guided in-Vivo Needle-Based Confocal Laser Endomicroscopy in the Prostate: Safety and Feasibility Study in 2 Patients. Technol Cancer Res Treat. 2022 Jan-Dec;21:15330338221093149. doi: 10.1177/15330338221093149. PMID 35790459
- [Derived] Swaan A, Mannaerts CK, Scheltema MJ, Nieuwenhuijzen JA, Savci-Heijink CD, de la Rosette JJ, van Moorselaar RJA, van Leeuwen TG, de Reijke TM, de Bruin DM. Confocal Laser Endomicroscopy and Optical Coherence Tomography for the Diagnosis of Prostate Cancer: A Needle-Based, In Vivo Feasibility Study Protocol (IDEAL Phase 2A). JMIR Res Protoc. 2018 May 21;7(5):e132. doi: 10.2196/resprot.9813. PMID 29784633